CLINICAL TRIAL: NCT00081523
Title: Studies of the Natural History of Sickle Cell Disease
Brief Title: Natural History of Sickle Cell Disease
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040161; 04-H-0161
Record Dates: First submitted 2004-04-15; First posted 2004-04-15 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01-02

CONDITIONS: Pain Crisis
Keywords: Hemoglobin; Acute Chest Syndrome; Treatment Options; Nitric Oxide; Pulmonary Hypertension; Natural History
MeSH Terms: conditions — Acute Chest Syndrome; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Individuals with known or suspected sickle cell disease

SUMMARY:
This study is not a treatment protocol and no experimental treatments are involved. Study participants may be seen as needed for clinical, translational and basic research studies, or as medically indicated. Subjects will receive their general medical care outside the NIH and will be seen at our clinic or at CNHS with varying frequency. Subjects may be seen for multiple visits. Subjects may be asked to return for additional testing as needed. Clinical care for patients with sickle cell disease will be provided as appropriate through the Sickle Cell Clinic and the inpatient clinical center....

DETAILED DESCRIPTION:
This protocol will permit the establishment of a repository of biospecimens from individuals affected with sickle cell disease to identify and evaluate underlying disease mechanism(s), and to facilitate understanding of the pathogenesis and natural history of vaso-occlusive painful crisis and other complications of the disease. Patients will be evaluated with a medical history and physical examination and routine laboratory studies will be obtained as needed to assess diagnosis, disease activity, and disease complications and to monitor for treatment-related responses and toxicities. This protocol may also provide for the continued storage and analysis of clinical and research data, and biospecimens previously obtained from other NIH Institutional Review Board (IRB)-approved protocols with subject consent.

Patients eligible for other research protocols will be offered an opportunity to participate in these studies after signed informed consent has been obtained. Apart from such protocols, any medical care or additional tests/investigations recommended or provided to the patient will be consistent with routine standards of practice and will be provided in consultation with the patient s referring physician.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals with known or suspected sickle cell disease
* 2 years of age and older
* Willing to provide informed consent or appropriate informed consent from parent or legal guardian
* Patients seen at sickle outpatient clinics at any one of the participating centers (CNHS or NIH).

EXCLUSION CRITERIA:

* Patient and/or guardian unable and unwilling to give informed consent or assent.
* Patients less than 2 years of age.

Individuals with known or suspected sickle cell disease will meet the inclusion criteria to enroll in this protocol and can undergo study activities. However, if the individual is found not to have sickle cell disease after enrollment, they will be removed from the protocol, and their research samples will be discarded but they will be counted toward the study accrual. The study team will notify the individual about their removal from the study and explain the reason for it. Any necessary regulatory reporting will also be completed.

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be open to all eligible subjects based on inclusion and exclusion criteria and who provide informed consent. Patients may self-refer, be recruited through the NIH office of recruitment, and may include patients participating on other NIH IRB approved protocols. The study will also be open to all eligible pediatric patients receiving medical care for SCD at Children s National.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2004-04-29 (Actual)

PRIMARY OUTCOMES:
To gather, through clinical experience, information regarding the natural history, co-morbid conditions and outcomes, and complications relating to sickle cell disease and other hemolytic disorders in minority/ethnic patients | ongoing
  Better characterization of the natural history of sickle cell disease

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (3):
- United States (3):
  - Childrens National Health Center, Washington D.C., District of Columbia
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
The team is in the process of making a determination.

REFERENCES:
- [Derived] Parrow NL, Doherty JM, Conrey A, Thein SL, Fleming RE. Relationships Between Markers of Iron Status and Hematological Parameters in Patients With Sickle Cell Disease. Adv Hematol. 2024 Dec 3;2024:9872440. doi: 10.1155/ah/9872440. eCollection 2024. PMID 39659429
- [Derived] Tumburu L, Ghosh-Choudhary S, Seifuddin FT, Barbu EA, Yang S, Ahmad MM, Wilkins LHW, Tunc I, Sivakumar I, Nichols JS, Dagur PK, Yang S, Almeida LEF, Quezado ZMN, Combs CA, Lindberg E, Bleck CKE, Zhu J, Shet AS, Chung JH, Pirooznia M, Thein SL. Circulating mitochondrial DNA is a proinflammatory DAMP in sickle cell disease. Blood. 2021 Jun 3;137(22):3116-3126. doi: 10.1182/blood.2020009063. PMID 33661274
- [Derived] Giudice V, Feng X, Lin Z, Hu W, Zhang F, Qiao W, Ibanez MDPF, Rios O, Young NS. Deep sequencing and flow cytometric characterization of expanded effector memory CD8+CD57+ T cells frequently reveals T-cell receptor Vbeta oligoclonality and CDR3 homology in acquired aplastic anemia. Haematologica. 2018 May;103(5):759-769. doi: 10.3324/haematol.2017.176701. Epub 2018 Feb 1. PMID 29419434
- [Derived] Nguyen KL, Tian X, Alam S, Mehari A, Leung SW, Seamon C, Allen D, Minniti CP, Sachdev V, Arai AE, Kato GJ. Elevated transpulmonary gradient and cardiac magnetic resonance-derived right ventricular remodeling predict poor outcomes in sickle cell disease. Haematologica. 2016 Feb;101(2):e40-3. doi: 10.3324/haematol.2015.125229. Epub 2015 Nov 20. No abstract available. PMID 26589907
- [Derived] Wang X, Mendelsohn L, Rogers H, Leitman S, Raghavachari N, Yang Y, Yau YY, Tallack M, Perkins A, Taylor JG 6th, Noguchi CT, Kato GJ. Heme-bound iron activates placenta growth factor in erythroid cells via erythroid Kruppel-like factor. Blood. 2014 Aug 7;124(6):946-54. doi: 10.1182/blood-2013-11-539718. Epub 2014 Jun 10. PMID 24916507
- [Derived] Koh C, Turner T, Zhao X, Minniti CP, Feld JJ, Simpson J, Demino M, Conrey AK, Jackson MJ, Seamon C, Kleiner DE, Kato GJ, Heller T. Liver stiffness increases acutely during sickle cell vaso-occlusive crisis. Am J Hematol. 2013 Nov;88(11):E250-4. doi: 10.1002/ajh.23532. Epub 2013 Aug 1. PMID 23828202
- [Derived] Tumblin A, Tailor A, Hoehn GT, Mack AK, Mendelsohn L, Freeman L, Xu X, Remaley AT, Munson PJ, Suffredini AF, Kato GJ. Apolipoprotein A-I and serum amyloid A plasma levels are biomarkers of acute painful episodes in patients with sickle cell disease. Haematologica. 2010 Sep;95(9):1467-72. doi: 10.3324/haematol.2009.018044. Epub 2010 Apr 7. PMID 20378559
- [Derived] Olnes M, Chi A, Haney C, May R, Minniti C, Taylor J 6th, Kato GJ. Improvement in hemolysis and pulmonary arterial systolic pressure in adult patients with sickle cell disease during treatment with hydroxyurea. Am J Hematol. 2009 Aug;84(8):530-32. doi: 10.1002/ajh.21446. PMID 19536844
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2004-H-0161.html